CLINICAL TRIAL: NCT00886249
Title: Depth of Focus Comparison Between Acrysof IQ and Acrysof Natural IOLs
Status: Withdrawn | Type: Observational
Why Stopped: The PI has determined not to continue the study.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Dr. Helga Sandoval, Medical University of South Carolina
Other Study IDs: HR#29924
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2009-10

CONDITIONS: Cataract; Vision
Keywords: Vision; Eye; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Acrysof IQ — Intraocular lens
  Other Names: Acrysof IQ SN60WF aspheric intraocular lens
Device: Acrysof Natural IOL — Intraocular Lens
  Other Names: Acrysof Natural SN60AT spherical IOL

SUMMARY:
The purpose of this study is to evaluate and compare the depth of focus and visual outcomes after implantation of the Acrysof IQ SN60WF aspheric intraocular lens (IOL) and the Acrysof Natural SN60AT spherical IOL.

DETAILED DESCRIPTION:
Cataract is prevalent throughout the world and IOLs are routinely implanted after the extraction of the cataractous lens. It is the most frequently performed surgery in the United States with an estimated 2-3 million procedures performed annually. With the aging population on the rise, as well as the increasing popularity of refractive intraocular lenses, the number of intraocular surgeries continues to rise.

Over the years, evolution of IOLs has broadened surgeon's armamentarium following cataract extraction. Traditionally spherical IOLs have been routinely implanted following cataract extraction for the correction of aphakia. Even though these IOLs improved the patient vision to 20/20 in most of the times, they did nott address the spherical aberration of the optical system.

Normally the cornea has a positive spherical aberration. Spherical aberration means that the light rays falling on the eye's periphery are either more (positive spherical aberration) or less (negative spherical aberration) refracted than the axial rays. Such aberration usually affects the functional vision of the patient such as contrast sensitivity, depth of focus (ability to see far, near and intermediate) and the perception of glare and haloes. Corneal spherical aberration is adequately neutralized by the negative spherical aberration of the crystalline lens until the age of 40. (1) When the cataractous lens is removed, the corneal spherical aberration is no longer neutralized and the optical system will have now a net positive spherical aberration.

Conventional IOLs implanted after phacoemulsification result in a spherical aberration of approximately 0.08 µm adding to the already positive corneal aberration of the eye. (2, 3) In order for the patient to reach the optimal functional vision, efforts have led to the development of the aspheric IOLs. Aspheric IOLs compensate for the positive spherical aberration of the cornea. They have been shown to improve the functional vision and optical quality in pseudophakic patients. (4, 5)

Acrysof IQ, an aspheric IOL was introduced after gaining FDA approval in May 2006. Its shares the basic design features of the Acrysof Natural IOL with the modifications of its optic design to acquire a posterior prolate surface reducing its central thickness. Unlike the cornea, it introduces negative spherical aberration (0.2 µm) that lowers the spherical aberration of the eye.(6) It has been reported to provide better contrast sensitivity, quality of vision and fewer aberration with the aspheric IOL compared to the conventional (spherical) IOL.(6,7,8) However, some studies have found that conventional (spherical) IOLs have better depth of focus than aspheric IOLs allowing the patient to achieve better intermediate and near vision.(5) Conversely, Mester et al found no difference in depth of focus between both IOLs.(7)

The purpose of this study is to evaluate and compare depth of focus and visual outcomes in eyes receiving the aspheric Acrysof IQ and those receiving the spherical Acrysof Natural IOL after routine cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

* Subject must have an age-related cataract in both eyes;
* Subject must be 40 years of age or older;
* Subject must desire cataract extraction;
* Expected maximum of 2 weeks and minimum of 1 week interval between the first and second eye surgeries; AND
* Subject must be willing and able to comply with scheduled visits and other study procedures.

Patient Exclusion Criteria:

* Preoperative ocular pathology: amblyopia, shallow anterior chamber, aniridia, history of iritis, iris neovascularization or iris atrophy, uveitis, medically uncontrolled glaucoma or advanced glaucomatous damage, rubella cataract, diabetic retinopathy, macular edema, retinal detachment, microphtalmus or macrophtalmus, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), etc.;
* Keratometric astigmatism exceeding 1.5 diopters;
* Uncontrolled diabetes;
* Use of any systemic or topical drug known to interfere with visual performance;
* Contact lens use during the active treatment portion of the trial;
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis;
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control;
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results;
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Prior history of eye surgery;
* Other ocular surgery at the time of the cataract extraction (except limbal relaxing incisions, LRI); OR
* History of trauma.

Surgical Exclusion Criteria:

The study lens should not be implanted and the patient should be excluded from the study if any of the following complications are encountered during surgery:

* Significant anterior chamber bleeding;
* Detached Descemet's membrane;
* Iris damage;
* Inability to achieve secure, symmetric, "in the bag" position of the IOL: posterior capsule rupture, radial tear in capsulorhexis, vitreous loss, zonular rupture; OR
* Use of corneal sutures for more than 1 week.

Post-implantation Exclusion Criteria:

* Haptic not in the capsular bag;
* Decentration of the IOL of more than 1.0 mm; OR
* Ocular pathologies potentially affecting visual acuity that were not evident prior to surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients of both sexes and any race undergoing routine bilateral phacoemulsification and intraocular lens implantation will be included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to evaluate and compare depth of focus and visual outcomes in eyes receiving the aspheric Acrysof IQ and those receiving the spherical Acrysof Natural IOL after routine cataract extraction. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Helga P Sandoval, MD, Principal Investigator — Associate Professor
Locations (1):
- Medical University of South Carolina, Storm Eye Institute, Charleston, South Carolina, United States